CLINICAL TRIAL: NCT07279064
Title: Comparison of Central Venous Pressure and Inferior Vena Cava Distensibility Index in Assessing Fluid Responsiveness in Septic Shocked Patients
Brief Title: Central Venous Pressure Versus Inferior Vena Cava Distensibility Index in Assessing Fluid Responsiveness in Septic Shocked Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa Abdelmomen Helal, Comparison of Central venous pressure and Inferior vena cava distensibility index in assessing fluid responsiveness in septic shocked patients, Assiut University
Other Study IDs: CVP-IVCDI-IN SEPTIC SHOCK
Record Dates: First submitted 2025-09-30; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-11

CONDITIONS: Central Venous Pressure and Inferior Vena Cava Distensibility Index in Assessing Fluid Responsiveness in Septic Shocked Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Ultrasound guided inferior vena cava distensibility index — This intervention involves bedside ultrasound measurement of the inferior vena cava (IVC) diameter and calculation of the IVC distensibility index. Assessments will be performed both at initial presentation and after fluid resuscitation in shock patients. The procedure is non-invasive, rapid, and performed according to standardized emergency ultrasound protocols.

SUMMARY:
This study aims to compare ultrasound-guided inferior vena cava distensibility index(IVC_DI) assessment with central venous pressure (CVP) monitoring for the detection of hypovolemia in septic shocked patients in the emergency department. The primary objective is to evaluate the diagnostic accuracy and clinical utility of IVC distinsisibility index compared to CVP values in both early and post- resuscitation phases. The study will prospectively enroll septic shocked patients, collect demographic and clinical data, and analyze the correlation between IVC DI and CVP measurements to determine their role in guiding fluid resuscitation and hemodynamic management

DETAILED DESCRIPTION:
Sepsis and septic shock remain among the leading causes of morbidity and mortality in intensive care units worldwide. Septic shock is defined as a subset of sepsis characterized by profound circulatory, cellular, and metabolic dysfunction, associated with a high risk of death despite adequate fluid resuscitation, vasopressor support, and infection source control. The cornerstone of early septic shock management is hemodynamic resuscitation, with intravenous fluids serving as the first-line therapy to restore effective circulating blood volume, improve cardiac output, and optimize tissue perfusion. However, while adequate fluid administration is lifesaving, excessive fluid loading can be detrimental, leading to interstitial edema, impaired oxygen delivery, increased intra-abdominal pressure, and pulmonary edema that may worsen outcomes. Therefore, precise identification of patients who are "fluid responsive" is of paramount clinical importance.

A direct comparison between CVP (as a traditional, static marker) and IVC distensibility index (as a dynamic marker) in patients with septic shock is essential to determine their relative value in guiding fluid resuscitation. This study aims to evaluate and compare the predictive accuracy, feasibility, and clinical applicability of these two parameters as tools for identifying fluid responsiveness in septic shock patients. The results may provide valuable insight into optimizing fluid resuscitation strategies, minimizing fluid overload, and ultimately improving patient outcomes.

ELIGIBILITY:
1. Inclusion criteria:

   * Adult patients (≥18 years old) both gender. with a clinical diagnosis of septic shock according to Sepsis-3 criteria (persistent hypotension require vasopressors to maintain MAP ≥65 mmHg and serum lactate >2 mmol/L despite adequate fluid resuscitation).(2,3).
   * with a central venous catheter in place for CVP monitoring. .awho require fluid resuscitation.
2. Exclusion criteria:

.pregnant patients. .Patients with significant right heart failure or severe tricuspid regurgitation (5)..

.Patients with increased intra-abdominal pressure or conditions affecting IVC diameter (9).

.Patients with arrhythmias (e.g., atrial fibrillation) that interfere with preload assessment (6).

.Patients who refuse participation.

* patients with contraindications to cvp (coagulopathy,distortion in anatomy of neck,....)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will include adult patients aged (≥18 years old) yearpresenting with septic shock to the emergency department and requiring volume status assessment through both IVC ultrasound and central venous pressure monitoring
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
To compare the accuracy of Central Venous Pressure (CVP) and Inferior Vena Cava Distensibility Index (IVC-DI) in predicting fluid responsiveness in patients with septic shock. | All patients will have the measurements of CVP and IVC_DI on arrival within 30 min before resuscitation and after 60 min of resuscitation